CLINICAL TRIAL: NCT04931940
Title: The Effect of Higher Protein Dosing in Critically Ill Patients: A Multicenter Registry-based Randomized Trial - The EFFORT Trial and EFFORT Outcomes Sub-study
Brief Title: The EFFORT Trial and EFFORT Outcomes Sub-study (EFFORT-Outcomes)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Responsible Party: Principal Investigator, Daren K. Heyland, Director, Clinical Evaluation Research Unit at Kingston General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: The EFFORT Outcomes sub-study
Record Dates: First submitted 2021-05-31; First posted 2021-06-18 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Critical Illness; Malnutrition
MeSH Terms: conditions — Critical Illness; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Patients will receive a usual protein/amino acid dose (≤1.2 g/kg/d)
  Interventions: Dietary Supplement: Usual Care
- Higher Protein/Amino Acid Group (Active Comparator): Patients will receive a higher protein/amino acid dose (≥2.2 g/kg/d).
  Interventions: Dietary Supplement: Higher Protein/Amino Acid Group

INTERVENTIONS:
Dietary Supplement: Usual Care — Patients will receive the usual protein dosage at ≤1.2 g/kg/day for up to 28 days in the ICU
  Arms: Usual Care
Dietary Supplement: Higher Protein/Amino Acid Group — Patients will receive high protein dosage at ≥2.2 g/kg/day for up to 28 days in the ICU
  Arms: Higher Protein/Amino Acid Group

SUMMARY:
The investigators will evaluate the effects of higher protein/amino acid dosing (≥2.2 g/kg/d) vs usual care of protein/amino acid dosing (≤1.2 g/kg/d) over muscle mass in nutritionally high risk ill patients

DETAILED DESCRIPTION:
The EFFORT Outcomes is a sub-study of the parent EFFORT trial; a multi-center, pragmatic, volunteer-driven, registry-based, randomized, clinical trial of 4000 nutritionally high-risk critically ill patients in the intensive care unit. Patients will be randomized to 1 of 2 treatment groups: a usual care prescription (≤1.2 g/kg/d) or a higher prescription (≥2.2 g/kg/d) of protein. Other than the protein amount the patient is randomized to, the remainder of care provided to randomized patient will be at the discretion of ICU providers. In both groups, targets will be achieved through any combination of enteral nutrition (high protein content in high group if available), protein supplements, and parenteral nutrition or amino acids only (as clinically available). The only difference between the 2 groups is the protein targets that are set. Similar efforts should be used in both groups to achieve at least 80% of these targets. The remainder of care provided to eligible patients will be at the discretion of ICU providers.

In patients included in the OUTCOMES sub-study, we will test the patient's functional recovery and long-term quality of life. Patients will undergo the US measures at baseline (within 24 hours of randomization, 10 days post randomization (if still in hospital) and just prior to hospital discharge. In the event that hospital discharge is prior to day 10, the day 10 measure will not be done. To ensure standardization and quality in the measures, we have created high quality training materials and will have US films sent centrally to abstract all measurements. In the first 10 patients enrolled in the US sub-study, participating sites will conduct a run-in phase where their submitted data will be evaluated for quality and reliability (both intra and inter-rater reliability) to ensure subsequent measures are of high quality. Nutritional and clinical data for these patients will be included in the parent EFFORT trial but the US measures may be omitted if quality is poor.

The investigator has posed the following research question:

Primary Outcome of the OUTCOMES Sub-study

The primary outcome will be the walking distance achieved during a 6-minute walk test (6MWT) measured at hospital discharge. Implementation of the test will be based upon the 2014 ATS standards, with adaptation, as needed, for the in-patient setting and ICU survivor population. The 6MWT is a reliable, valid, responsive measure of physical function for survivors of acute respiratory failure.

Secondary measures for this OUTCOMES sub-study will include;

1. Overall strength using Medical Research Council (MRC) sum-score evaluated via standardized "manual muscle testing" with each of 12 muscle groups assessed using a 6-point MRC scale and summed to a total score (range: 0-60).
2. Quadriceps force, via hand-held dynamometry (HHD) for of both lower extremities. Each will be scored by, averaging the results of 3 trials.
3. Distal strength measured via isometric handgrip strength via a hydraulic hand dynamometer performed bilaterally as per American Society of Hand Therapist guidelines and evaluated using normal values.
4. Short Physical Performance Battery (SPPB) which measures balance, walking speed and rising from a chair
5. Functional Status Score for ICU (FSS-ICU), which is a 5-item, 35-point assessment of bed mobility, transfers, and ambulation. designed for ICU patients, and was designed and validated specifically in ICU patients evaluated 8-point Functional Independence Measure (FIM) response scale used throughout rehabilitation assessments, and is responsive to change during recovery for ICU patients.

Lastly, outcomes after hospital discharge will be assessed via 6-month phone-based follow-up. Health-related quality of life (QOL) will be measured using SF-36 version 2 (SF-36 v2) and EQ-5D-5L. The SF-36 is valid and reliable across a variety of patient groups, including ICU survivors. The EQ-5D-5L is included, in addition to SF-36 v2, because it is suitable for patients with inattention and fatigue, recommended for use in ICU survivors. Physical functional status will be measured using Katz activities of daily living (ADL) and Lawton's Instrumental ADL (IADL). In order to improve retention, a call will be made to participants at 3 months to update contact information and act as a reminder of upcoming follow-up assessments to be completed at the 6-month time point.

Overall Hypothesis: Compared to receiving a lower dose of protein/amino acids, the administration of a higher dose of protein/amino acids (a consequence of having a higher prescription) to nutritionally high-risk critically ill patients will be associated with greater muscle mass, improved survival and a quicker rate of recovery.

ELIGIBILITY:
Inclusion Criteria:

1. - ≥18 years old
2. - Nutritionally 'high-risk' (meeting one of the below criteria)

   1. Low (≤25) or High BMI (≥35)
   2. Moderate to severe malnutrition (as defined by local assessments). We will document the means by which sites are making this determination and capture the elements of the assessment (history of weight loss, history of reduced oral intake, etc.).
   3. Frailty (Clinical Frailty Scale 5 or more from proxy)
   4. Sarcopenia- (SARC-F score of 4 or more from proxy)
   5. From point of screening, projected duration of mechanical ventilation >4 days
3. - Requiring mechanical ventilation with actual or expected total duration of mechanical ventilation >48 hours

Exclusion Criteria:

1. >96 continuous hours of mechanical ventilation before screening
2. Expected death or withdrawal of life-sustaining treatments within 7 days from screening
3. Pregnant
4. The responsible clinician feels that the patient either needs low or high protein
5. Patient requires parenteral nutrition only and site does not have products to reach the high protein dose group.
6. Not ambulating independently prior to illness that leads to ICU admission (use of gait aid permitted)
7. Lower extremity injury or impairments that prevents them from walking prior to hospital discharge (e.g. amputation, knee/hip injury)
8. Pre-existing cognitive impairment or language barrier that prohibits outcomes assessment
9. Pre-existing primary severe systemic neuromuscular disease resulting in severe weakness pre-ICU (e.g., Guillain Barre) 10 Intracranial or spinal process affecting motor function

11. Patients in hospital >5 days prior to ICU admission 12. Not expected to stay ≥4 days after enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test (6MWT) | Within 72 hours before discharge from the hospital
  walking distance achieved during a 6-minute walk test (6MWT) measured at hospital discharge

SECONDARY OUTCOMES:
Quadriceps Muscle Mass | Day 1 and Day 10 of randomization, and within 72 hours before discharge from the hospital
  Quadriceps muscle thickness and cross-sectional area measured by ultrasonography
Functional Status Score for ICU (FSS-ICU) | Day 1 of randomization (surrogate interview), within 72 hours before discharge from the ICU and hospital (by trained physiotherapist)
  which is a 5-item, 35-point assessment of bed mobility, transfers, and ambulation. designed for ICU patients, and was designed and validated specifically in ICU patients evaluated 8-point Functional Independence Measure (FIM) response scale used throughout rehabilitation assessments, and is responsive to change during recovery for ICU patients
Handgrip strength | Within 72 hours before discharge from the ICU and hospital
  measured via isometric hand grip strength via a hydraulic hand dynamometer performed bilaterally as per American Society of Hand Therapist guidelines and evaluated using normal values.
Short Physical Performance Battery (SPPB) | Within 72 hours before discharge from the ICU and hospital
  which measures balance, walking speed, and rising from a chair
Quadriceps force | Within 72 hours before discharge from the hospital
  via hand-held dynamometry (HHD) for of both lower extremities. Each will be scored by, averaging the results of 3 trials.
Overall strength | Within 72 hours before discharge from the hospital
  using Medical Research Council (MRC) sum-score evaluated via standardized "manual muscle testing" with each of 12 muscle groups assessed using a 6-point MRC scale and summed to a total score (range: 0-60)

OTHER OUTCOMES:
Health related quality of life by Short-Form 36 version 2 (SF-36 v2) | 6 months post-randomization
  The SF-36 physical function domain ranges from 0-100. Higher scores indicate better outcome.
Health-related Quality of life by Euro Quality of Life 5 Dimension 5 level (EQ-5D-5L) | 6 months post-randomization
  The overall health scale where the rater selects a number between 1-100 to describe the condition of their health, 100 being the best imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Daren K Heyland, DM, Principal Investigator — Clinical Evaluation Research Unit
Locations (2):
- Gold Coast Hospital and Health Service, Gold Coast, Australia
- University of Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided